CLINICAL TRIAL: NCT04637763
Title: A Phase 1, Multicenter, Open-Label Study of CB-010, a CRISPR-Edited Allogeneic Anti-CD19 CAR-T Cell Therapy in Patients With Relapsed/Refractory B Cell Non-Hodgkin Lymphoma (ANTLER)
Brief Title: CRISPR-Edited Allogeneic Anti-CD19 CAR-T Cell Therapy for Relapsed/Refractory B Cell Non-Hodgkin Lymphoma (ANTLER)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Caribou Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB10A
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma, Non-Hodgkin; Relapsed Non Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Non Hodgkin Lymphoma; Lymphoma; B Cell Lymphoma; B Cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: The CB10A clinical study consists of (Part A) 3 + 3 design with three dose levels.
  (Part B) Expansion portion patients will receive CB-010 at the dose determined in Part A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation of CB-010 (Experimental): Patients with relapsed or refractory non-Hodgkin lymphoma will receive CB-010 following lymphodepletion.
  Interventions: Genetic: CB-010; Drug: Cyclophosphamide; Drug: Fludarabine
- Expansion of CB-010 (Experimental): Patients with relapsed or refractory non-Hodgkin lymphoma will receive CB-010 following lymphodepletion.
  Interventions: Genetic: CB-010; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Genetic: CB-010 — CB-010 is a CRISPR-edited allogeneic CAR-T cell therapy targeting CD19.
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion
Drug: Fludarabine — Chemotherapy for lymphodepletion

SUMMARY:
CB010A is a study evaluating safety, emerging efficacy, pharmacokinetics and immunogenicity of CB-010 in adults with relapsed/refractory B cell non-Hodgkin lymphoma after lymphodepletion consisting of cyclophosphamide and fludarabine.

DETAILED DESCRIPTION:
This clinical trial is a first-in-human, Phase 1, multicenter, open-label evaluation of safety and emerging efficacy of CB-010 in adults with relapsed/refractory B cell non-Hodgkin lymphoma. The study is conducted in two parts: Part A is dose escalation following a 3 + 3 design, with sequential, prespecified, increasing doses. Part B is the expansion portion where patients will receive CB-010 at the dose determined in Part A.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 at the time of enrollment
* Documented diagnosis of relapsed or refractory non-Hodgkin lymphoma after prior standard of care
* Eastern Cooperative Oncology Group performance status 0 or 1
* Adequate hematologic, renal, liver, cardiac and pulmonary organ function

Exclusion Criteria:

* Prior therapy with an anti-CD19 targeting agent
* Active or chronic graft versus host disease requiring therapy
* Prior allogeneic stem cell transplantation
* Central nervous system (CNS) lymphoma, prior CNS malignancy
* Prior seizure disorder, cerebrovascular ischemia, dementia, cerebellar disease or autoimmune disease with CNS involvement.
* Primary immunodeficiency
* Current or expected need for systemic corticosteroid therapy
* Current thyroid disorder. Hypothyroidism controlled with stable hormone replacement is permitted
* Other malignancy within 2 years of study entry, except curatively treated malignancies or malignancies with low risk of recurrence
* Unwillingness to follow extended safety monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures number of patients with dose-limiting toxicities (Part A). | 28 days following CB-010 infusion
  Incidence of adverse events defined as dose-limiting toxicities with onset within 28 days after CB-010 infusion.
Primary outcome evaluates tumor response (Part B) | Up to 12 months
  The primary endpoint is objective response rate.

CONTACTS AND LOCATIONS:
Locations (38):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - HonorHealth, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Chao Family Comprehensive Cancer Center/University of California Irvine, Orange, California
  - Advent Health, Orlando, Florida
  - Bone and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Holden Comprehensive Cancer Center at the University of Iowa, Iowa City, Iowa
  - University of Kentucky Markey Cancer, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Hackensack Medical Center, Hackensack, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - Nyu Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Ohio State University James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University (VCU), Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - Epworth Healthcare, Richmond, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Israel (4):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Medical Center, Tel Aviv
  - The Sheba Fund for Health Services and Research (R.A.), Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Undecided